CLINICAL TRIAL: NCT06215677
Title: Efficacy of Neoadjuvant Immunotherapy for T4 Deficient Mismatch Repair (dMMR) Colon Cancer: A Prospective, Single-arm, Phase Ⅱ Clinical Trial
Brief Title: Neoadjuvant Immunotherapy for T4 dMMR Colon Cancer
Acronym: NITDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, XIAO Yi, MD, Director, Head of Colorectal surgery, Principal Investigator, Clinical Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K5121
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer; Mismatch Repair Deficiency; Immunotherapy
MeSH Terms: conditions — Colonic Neoplasms; Turcot syndrome | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant immunotherapy (Experimental)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg for 3 cycles. Patients will undergo surgery 2-3 weeks after the last cycle of immunotherapy, type and extent of the surgery will be selected by the surgeon.

SUMMARY:
Due to dMMR colon cancer patients respond poorly to conventional chemotherapy, but immunotherapy can significantly improve the pCR in this group of patients, this study intends to explore whether neoadjuvant immunotherapy can improve the R0 resection rate with preservation of adjacent organs in T4 colon cancer patients with dMMR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. ECOG score 0-2;
3. Adenocarcinoma confirmed by pathology and dMMR confirmed by IHC or PCR;
4. Tumor located in cecum, ascending colon, transverse colon and sigmoid colon;
5. Patients with clinical stage cT4: (1) Loss of space between tumor and adjacent organs or invasion of adjacent organs as assessed by enhanced CT; (2) R0 resection cannot achieve according to intraoperative exploration;
6. No evidence of distant metastasis;
7. Newly treated patients who have not received treatment including chemotherapy and surgery;
8. Liver, kidney and other organs have good function and can tolerate chemotherapy and surgery;
9. Patients and family members can understand the study protocol, voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

1. A history of other malignant tumors (other than cured basal cell carcinoma, cervical carcinoma in situ, surgically treated localized prostate cancer, or surgically resected breast ductal carcinoma in situ) within the past 5 years;
2. Complicated with intestinal obstruction, intestinal perforation, gastrointestinal bleeding and other patients requiring emergency surgery; pregnant or lactating women;
3. Patients with a history of severe mental illness, immune disease, hormone medication;
4. Patients contraindicated by immunotherapy or surgery;
5. Participated in other clinical researchers in the past 3 months;
6. Any other circumstances that the investigator considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2030-02-10 (Estimated)

PRIMARY OUTCOMES:
the rate of R0 resection | Tumour specimen evaluated within 2 weeks after surgery
  No tumor infiltration within 1 mm of the surgical margins

SECONDARY OUTCOMES:
Pathological complete response (pCR) | Tumour specimen evaluated within 2 weeks after surgery.
  Number of patients with pCR evaluated according to the Mandard tumour regression grading system
diesease-free survival | 3 years
  No tumor regrowth or recurrence or metastasis found
overall survival | 5 years
  Refers to the proportion of patients still alive at 5 years after surgery
Safety and tolerability of Camrelizumab administered | Up to approximately 9 weeks
  Determined by the incidence and severity of treatment related adverse events according to CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing